CLINICAL TRIAL: NCT03477253
Title: Laparoscopic Cholecystectomy for Management of Acute Calculous Cholecystitis Within Versus After 3 Days of Disease Onset
Brief Title: Laparoscopic Cholecystectomy in Management of ACC Within Versus After 3 Days
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Elmahdy Ali Abdel Rahman Morsy, Resident Doctor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC in management of ACC
Record Dates: First submitted 2018-03-14; First posted 2018-03-26 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Acute Calculous Cholecystitis
Keywords: Acute calculous cholecystitis; Laparoscopic cholecystectomy; Early laparoscopic cholecystectomy; Late laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: 62 patients with acute calcular cholecystitis are divided into 2 study groups by the time of laparoscopic cholecystectomy comparing to onset of symptoms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC within 72 hours of disease onset (Active Comparator): Immediate laparoscopic cholecystectomy within 72 hours of the onset of symptoms was performed in these patients
  Interventions: Procedure: Laparoscopic cholecystectomy
- LC after 72 hours of disease onset (Active Comparator): Late laparoscopic cholecystectomy after 72 hours of the onset of symptoms was performed in these patients
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — The use of laparoscopic cholecystectomy in management of acute calculous cholecysitits

SUMMARY:
This study was aimed to assess the outcome of laparoscopic cholecystectomy in acute calculous cholecystitis in terms of conversion rates, postoperative complications and length of hospital stay within and after 3 days of symptoms onset.

DETAILED DESCRIPTION:
The study aims to evaluate the safety and competency of laparoscopic cholecystectomy as surgical management of acute calculous cholecystitis within and after 72h of symptom onset.

This study included 62 patients with acute calculous cholecystitis. Patients are divided into 2 study groups by the time of laparoscopic cholecystectomy comparing to the onset of symptoms and categorized as Group A & B. Immediate laparoscopic cholecystectomy is performed in Group A. while late laparoscopic cholecystectomy is performed in Group B. Patients in both groups monitored since admission, during operations, and along the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal pain characteristic of Acute Cholecystitis, Positive Murphy's sign, Total Leucocyte Count > 10,000/ uL, and (4) Ultra-sonographic evidence of Acute Calculous Cholecystitis.
2. Initial surgical management planned for immediate laparoscopic cholecystectomy.
3. Patients who are fit for laparoscopy and general anesthesia.
4. Patient who agree to provide short term outcome data and agree to provide contact information.

Exclusion Criteria:

1. Patients with ultra-sonographic findings of common bile duct calculi, pancreatitis, gall bladder perforation, gall bladder gangrene or gall bladder abscess.
2. Patients with other associated abdominal pathology.
3. Patients with any previous abdominal surgery or any significant systemic disease.
4. Septic shock.
5. Pregnancy/ Breast-feeding mothers.
6. Participation in an additional drug or device study and inability to offer informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Comparison between early and late laparoscopic cholecystectomy regarding Operation time | intra-operative
  comparing the needed intra-operative time for laparoscopic cholecystectomy within and after 3 days of the onset of acute calcular cholecystitis , time will be measured by minutes
Comparison between early and late laparoscopic cholecystectomy regarding difficulty of operation | intra-operative
  comparing the difficulty of laparoscopic cholecystectomy within and after 3 days of the onset of acute calculous cholecystitis, difficulty will be assessed by the rate of conversion to open cholecystectomy
comparison between early and late laparoscopic cholecystectomy regarding post operative pain | within 1month post operative
  comparing between laparoscopic cholecystectomy within and after 3 days of the onset of acute cholecystitis regarding the presence and duration of post operative pain , pain will be measured by either the pain responded to regular NSAIDs or needed the administration of narcotics
Duration of postoperative hospital stay | within 2 weeks post-operative
  comparing post-operative duration of hospital stay after laparoscopic cholecystectomy within and after 3 days of the onset of acute calcular cholecystitis ,duration will be measured by post operative days spent in the hospital

SECONDARY OUTCOMES:
comparison between early and late laparoscopic cholecystectomy regarding post operative bile leakage | first 72 hours post-operative
  compare between laparoscopic cholecystectomy within and after 3 days of the onset of acute cholecystitis regarding the presence and amount of bile leakage
comparison between early and late laparoscopic cholecystectomy regarding post operative bleeding | 7 days postoperative
  compare between laparoscopic cholecystectomy within and after 3 days of the onset of acute cholecystitis regarding the presence and amount of postoperative bleeding
presence of any wound complication by examining the wound | within 10 days post-operative
  comparison between early and late laparoscopic cholecystectomy concerning the presence and rate of wound infection by clinical examination post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elmahdy, Study Chair — Assiut University; Gamal Abdel Hameed, Study Director — Assiut University; Gamal Makhlouf, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Yuval JB, Mizrahi I, Mazeh H, Weiss DJ, Almogy G, Bala M, Kuchuk E, Siam B, Simanovsky N, Eid A, Pikarsky AJ. Delayed Laparoscopic Cholecystectomy for Acute Calculous Cholecystitis: Is it Time for a Change? World J Surg. 2017 Jul;41(7):1762-1768. doi: 10.1007/s00268-017-3928-4. PMID 28251270
- [Background] Gomes CA, Junior CS, Di Saverio S, Sartelli M, Kelly MD, Gomes CC, Gomes FC, Correa LD, Alves CB, Guimaraes SF. Acute calculous cholecystitis: Review of current best practices. World J Gastrointest Surg. 2017 May 27;9(5):118-126. doi: 10.4240/wjgs.v9.i5.118. PMID 28603584
- [Background] Terho PM, Leppaniemi AK, Mentula PJ. Laparoscopic cholecystectomy for acute calculous cholecystitis: a retrospective study assessing risk factors for conversion and complications. World J Emerg Surg. 2016 Nov 16;11:54. doi: 10.1186/s13017-016-0111-4. eCollection 2016. PMID 27891173
- [Background] Bagla P, Sarria JC, Riall TS. Management of acute cholecystitis. Curr Opin Infect Dis. 2016 Oct;29(5):508-13. doi: 10.1097/QCO.0000000000000297. PMID 27429137
- [Background] Dudchenko MO, Kravtsiv MI, Lyulka MO, Lyakhovsky VI, Furman DD, Bondar LD. [TREATMENT OF ACUTE CALCULOUS CHOLECYSTITIS: "EARLY" OR "PLANNED" LAPAROSCOPIC CHOLECYSTECTMIVY]. Klin Khir. 2015 Jun;(6):19-21. Ukrainian. PMID 26521459
- [Background] Polo M, Duclos A, Polazzi S, Payet C, Lifante JC, Cotte E, Barth X, Glehen O, Passot G. Acute Cholecystitis-Optimal Timing for Early Cholecystectomy: a French Nationwide Study. J Gastrointest Surg. 2015 Nov;19(11):2003-10. doi: 10.1007/s11605-015-2909-x. Epub 2015 Aug 12. PMID 26264362